CLINICAL TRIAL: NCT06557486
Title: The Effects of Mindfulness-Based Stress Reduction Program on the Psychological and Physiological Stress of Family or Caregivers of Children With Motor Disabilities Due to a Neurological Disorder: A Randomized Controlled Trial
Brief Title: The Effects of Mindfulness-Based Stress Reduction Program for Family or Caregivers of Children With Motor Disabilities
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, Clàudia Arumí, Principal Investigator, Universitat de Lleida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ULleida2
Record Dates: First submitted 2024-07-30; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Stress, Psychological; Stress, Emotional; Stress
MeSH Terms: conditions — Stress, Psychological | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Stress reduction arm (Experimental)
  Interventions: Behavioral: Mindfulness-Based Stress reduction
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress reduction — Participants assigned to the 8-week mindfulness program attended weekly 120-150 minute in-person group sessions for the entire duration. In these sessions, the instructor progressively will introduce and guide formal mindfulness practices while facilitating the sharing of experiences.
  Arms: Mindfulness-Based Stress reduction arm

SUMMARY:
The present study aims to investigate the effect of a mindfulness-based program on perceived stress, severity of anxiety, parents'/caregivers' quality of life and their children, cortisol and IL-6 blood concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Not having attended previously a mindfulness course
* A score equal to or greater than 23 points at the PSS.
* >18 years old
* Children <18y with motor/physical disability due to a Neurological disorder.
* Spanish/Catalan speaking

Exclusion Criteria:

* Currently using drugs or any kind of medication related to stress, depression, anxiety or sleeping pills, such as steroid medicines.
* Regular meditation practice (once a week in the past 12 months)
* Diagnose of hypertension stage 2
* Pregnancy in the case of mothers
* Present hyperthyroidism
* Primary adrenal insufficiency syndromes such as Cushing syndrome or Addison disease
* Present any kind of infection or inflammation process, different from the interestingly to the present study that could differ the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress | baseline, two months (through study completion), and follow-up of one month
  To measure participants perceived stress, the Perceived Stress Scale 14 item Spanish version will be used (PSS 14). It consists of 14 items scored from 0 up to 4 (0=never, 1 = rarely 2= sometimes 3= usually 4 =almost always). The total scores on the scale can range from 0 (no stress) to 56 (extreme stress).
Cortisol levels | baseline and two months (through study completion)
  The cortisol measurement will be sampled with a serum blood test. It is recommended to advise the participants to be fasted. 63 Cortisol levels fluctuate throughout the day, being highest in the morning and lowest at night.63,64 The sample will be collected between 8-9 am to get the highest cortisol.

SECONDARY OUTCOMES:
Severity of clinic anxiety | baseline, two months (through study completion), and follow-up of one month
  To measure the severity of clinic anxiety, the Bech Anxiety Inventory will be used. It consists of 21 self-administered questions about how the individual has been feeling the last week, expressed in common anxiety symptoms. It takes up to 5-10 minutes. Scores 0-7 indicate minimal anxiety, 8-15 mild anxiety, 16-25 moderate anxiety and 26-63 severe anxiety. Each item on the BAI includes an anxiety symptom and for each of them, the participant must assess the degree to which they have been affected by it during the last week. Possible answers are: not at all, mildly but it didn't bother me much, moderately it wasn't pleasant at times, severely it bothered me a lot. (0 to 3 respectively).
Sleep Quality | baseline, two months (through study completion), and follow-up of one month
  To measure sleep quality, the Pittsburgh Sleep Quality Index (PSQI) will be assessed. It is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. The instrument should require between 5 and 10 min for completion. The questionnaire consists of a combination of Likert-type and open-ended questions (later converted to scaled scores using provided guidelines). Respondents are asked to indicate how frequently they have experienced certain sleep difficulties over the past month and to rate their overall sleep quality. Scores for each question range from 0 to 3, with higher scores indicating more acute sleep disturbances. Developers have suggested a cutoff score of 5 for the global scale. The seven component scores are then combined to produce a global PSQI score, which ranges from 0 to 21; higher scores reflect poorer sleep quality
Quality of Life assessment | baseline, two months (through study completion), and follow-up of one month
  To measure the impact of paediatric chronic health conditions on parents and the family, the last developed PedsQL™ Family Impact Module will be used. The module measures multidimensions parent self-report; physical, emotional, social, and cognitive functioning, communication, and worry. It is used to assess health-related QoL in children aged 2-18 years. It takes up to 5-10 minutes to be completed.It assesses 8 main factors: physical functioning (6 items), emotional functioning (5 items), social functioning (4 items), cognitive functioning (4 items), communication (3 items), worry (5 items), daily activities (3 items) and family relationships (5 items). The answers are given on a 5-point Likert scale (0 = it is never a problem, 4 = it is almost always a problem) and are reversed scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0) so that a greater score indicates better functioning
Blood pressure | baseline, two months (through study completion), and follow-up of one month
  BP will be measured, after 5 min of rest, three times at intervals of 1 minute using a sphygmomanometer. The clinical BP values used in the analysis will be the averages for the three measurements. BP measurements will be done pre-intervention, post-intervention and with a follow-up of one mont. both systolic and diastolic measures.
Resting Heart rate | baseline, two months (through study completion), and follow-up of one month
  HR will be measured, after 5 min of rest, three times at intervals of 1 minute using a pulsometer on the index finger. The clinical HR values used in the analysis will be the averages for the three measurements.
Respiratory rate | baseline, two months (through study completion), and follow-up of one month
  Respiratory rate will be measured after 5 min of rest, three times at intervals of 1 minute using the same sphygmomanometer of the BP. The clinical RR values used in the analysis will be the averages for the three measurements. RR measurements will be done pre-intervention, post-intervention and with a follow-up of one month.
Interleukin 6 (IL-6) | baseline and two months (through study completion)
  The same procedure will be taken for the IL-6 .65 Under homeostatic conditions, IL-6 levels in the circulation are as low as 1-5 pg/ml, but during inflammatory states, these levels can rise more than 1,000-fold

CONTACTS AND LOCATIONS:
Locations (1):
- Claudia Arumi, Lleida, Spain

IPD SHARING:
Plan to Share IPD: No